CLINICAL TRIAL: NCT06855186
Title: Symptom-Targeted Approach to Rehabilitation for Concussion (STAR-C): RCT of In-person vs Telehealth vs Wait List Control
Brief Title: Symptom-Targeted Approach to Rehabilitation for Concussion (STAR-C)
Acronym: STAR-C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); Tripler Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.2024.104d
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Mild Traumatic Brain Injury (mTBI)
Keywords: concussion; brain injury; cognitive rehabilitation; military; adults
MeSH Terms: conditions — Brain Concussion; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Treatment Waitlist (Other): Individuals randomized to this arm will go for 4 weeks without treatment. During this time, participants will be asked to remain stable on treatments that they are already receiving for their concussive symptoms; that is and should not start a new treatment or change their medication. At the end of the 4-week wait, participant's will be asked about any changes to treatments that they have received during this time, and participants will be asked to complete questionnaires. This visit can be complete in person or remotely. Participants will be randomized into the in-person or telemedicine group.
  Interventions: Behavioral: Symptom-Targeted Approach to Rehabilitation for Concussion
- In-Person STAR-C (Other): Individuals assigned to this treatment will receive in-person individual cognitive rehabilitation treatment conducted by credentialed speech or occupational therapists. Participants will complete up to three sessions per week (approximately 50 minutes each) for up to nine sessions plus one wrap up session. The treatment will include a focus on compensatory strategies and weekly homework assignments. Participants will work on personalized targets and assignments. The treatment will end with one wrap up session where participants will put together a plan for maintenance of what they have learned with their therapist's help.
  Interventions: Behavioral: Symptom-Targeted Approach to Rehabilitation for Concussion
- Telehealth STAR-C (Other): Individuals assigned to this treatment will receive individual cognitive rehabilitation treatment conducted by credentialed speech or occupational therapists via a telemedicine format. Participants will complete up to three sessions per week (approximately 50 minutes each) for up to nine sessions plus one wrap up session. The treatment will include a focus on compensatory strategies and weekly homework assignments. Participants will work on personalized targets and assignments. The treatment will end with one wrap up session where participants will put together a plan for maintenance of what they have learned with their therapist's help.
  Interventions: Behavioral: Symptom-Targeted Approach to Rehabilitation for Concussion

INTERVENTIONS:
Behavioral: Symptom-Targeted Approach to Rehabilitation for Concussion — This study is looking at a shortened version of a therapist-direct cognitive rehabilitation intervention, known as STAR-C. STAR-C is focused on strategy use, and for strategy use to become a habit the person must have the opportunity for high-dose spaced practice. Thus, in STAR-C each session includes opportunities for repeated practice and participants schedule practice times between sessions. Sometimes a new strategy requires learning new facts, in which case the clinician chooses ingredients such as self-quizzing or comparing and contrasting outcomes, which are effective for learning new facts and concepts.

SUMMARY:
Purpose: Investigators propose a three-arm RCT across two military treatment facilities:1) in-person STAR-C, 2) telehealth STAR-C, and 3) no treatment control. Outcomes will be assessed immediately and at one- and three-months post treatment.

Hypothesis/Objectives: STAR-C, delivered in-person and via telehealth, will be effective in decreasing everyday cognitive complaints among patients with a history of mTBI. Effectiveness will be moderated by patient characteristics. Stakeholder feedback will yield a process map for broad implementation of STAR-C in varied clinical environments.

DETAILED DESCRIPTION:
Specific Aim 1 (primary for RCT): To evaluate effectiveness of STAR-C.

Hypothesis 1a: In-Person STAR-C will lead to a greater decrease in everyday cognitive complaints (C4) compared to wait-list control.

Hypothesis 1b: Tele STAR-C will lead to a greater decrease in everyday cognitive complaints (C4) compared to wait-list control.

Specific Aim 2 (secondary): To evaluate maintenance of treatment effects using a practice based evidence approach.

Question 2a: What proportion of in-person STAR-C treatment effects (C4 and GAS) will be maintained at the 3-month follow-up?

Question 2b: What proportion of telehealth STAR-C treatment effects (C4 and GAS) will be maintained at the 3-month follow-up?

Specific Aim 3 (exploratory): To explore factors associated with heterogeneity in treatment response.

Question 3a: What factors prevented participants from achieving a ≥2-point improvement on the C4?

Question 3b: What factors prevented participants from maintaining ≥2-point improvement on the C4?

Question 3c: What factors prevented participants from achieving ≥2 out of 3 targets using GAS?

Question 3d: What factors contributed to participants maintaining or exceeding targets (GAS) at the 3-month follow-up?

Specific Aim 4 (implementation): Use stakeholder input (to include clinicians, administrators, and patients) from capacity assessment and after-action review to generate an implementation package for clinics interested in STAR-C.

Question 4: For what proportion of patients will clinicians rate STAR-C as acceptable, appropriate, and feasible (AIM/IAM/FIM)?

ELIGIBILITY:
Inclusion Criteria:

* mTBI defined per the VA/DoD Clinical Practice Guideline for the Management of Concussion-Mild Traumatic Brain Injury sustained in any context (deployment related or non-deployment-related) and at any time longer than 3 months previously.
* a score of 2, 3, or 4 on any of the four Cognitive items on the NSI, to include participants who have cognitive complaints.
* a score on the Word Reading Subtest of the Wide Range Achievement Test of a sixth-grade reading level or higher, to ensure participants can read study materials.

Exclusion Criteria:

* History of a moderate, severe, or penetrating TBI as defined by DoD/VA guidelines.
* Lifetime diagnosis of schizophrenia or other psychotic/thought disorder.
* Current participation in intensive behavioral health treatment (≥3 appointments /encounters per week) for any psychiatric or substance use disorder.
* Current participation in other treatments that target cognition within the last two weeks (i.e., healthcare provider-prescribed cognitive rehabilitation in a group or individual format of any time duration or involving digital/game-based format of more than 4 hours per week).
* History of a neurological disease affecting cognitive function, other than mild TBI, such as multiple sclerosis, stroke, brain tumor, or Parkinson Disease.
* Current, active suicidal or homicidal ideation.
* Daily use of narcotic pain medications.
* Lack of access to technology or internet/cell phone service that supports telemedicine.
* Current participation in other therapy targeting cognition (Note: This is not the same as Cognitive Behavioral Therapy/CBT which addresses psychological issues and may continue during participation in this research project).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 222 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Common Concussive Cognitive Complaints (C4) | From baseline to 3 months post treatment
  On the C4, patients are asked to "identify challenges that are new since your injury and affect your everyday functioning, so we can focus therapy on what is most important to you." For each question, the patient is asked to choose the number that shows how often this has caused problems for them in everyday life in the past two weeks. Responses are on a scale from 1 (not at all) to 5 (all the time). The reliability and validity of the C4 are acceptable (internal consistency of domains: 0.465 to 0.797; 4-week test-retest reliability of domains: 0.628 to 0.832; convergent validity with MMPI-3 Cognitive Complaints and Inefficiency scales and discriminant validity with MMPI-3 Activation and Eating Concerns scales).
Goal Attainment Scaling (GAS) | From treatment week 1 to 3 months post treatment
  As described above in the Summary of ongoing relevant clinical trials, in each session, the patient and therapist collaborate to identify a desired outcome for the patient's target and then scale it using a 5-point rating system. The patient's current state relative to the target is assigned a 0 on the scale, achievement of the desired target is +2, partial achievement is +1, and achievement beyond expectations is +3. Success is defined as a GAS score of 2 or 3.

SECONDARY OUTCOMES:
Evaluate maintenance of treatment effects | From baseline to 3 months post treatment
  Question 2a: At the 3-month follow-up, determine the proportion of in-person STAR-C participants with ≥2 points C4 improvement post treatment maintained their improvement using contingency table or McNemar test. Question 2b: At the 3-month follow-up, determine the proportion of telehealth STAR-C participants with ≥2 points C4 improvement post treatment maintained their improvement using contingency table or McNemar test. Question 2c: At the 1-month and 3-month follow-ups, describe rates of maintaining ≥2 points C4 improvement for the in-person and telehealth STAR-C groups.

OTHER OUTCOMES:
To explore factors associated with heterogeneity in treatment response. Statistical approach will be determined after potential factors are evaluated for differences between the RCT arms | From baseline to 3 months post treatment
  Question 3a: Determine what factors, if any, that may have prevented participants from achieving a ≥2 point C4 improvement at the end of treatment.
  Question 3b: Determine what factors, if any, that may have prevented participants from maintaining at ≥2 point C4 improvement at the 3-month follow-up. Question 3c: Determine what factors, if any, that may have prevented participants from achieving ≥2 out of 3 targets using GAS. Question 3d: Determine what factors, if any, that may have contributed to participants maintaining or exceeding targets (GAS) at the 3-month follow-up.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Desmond T. Doss Health Clinic, Wahiawa, Hawaii
  - Brooke Army Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Common Concussive Cognitive Complaints (C4); Goal Attainment Scaling (GAS); Audio recordings; Patient Characterization Measures (headache, sleep problems, dizziness, musculoskeletal injury and pain, medications, and use of commercial brain games); Neurobehavioral Symptom Inventory (NSI); Key Behaviors Change Inventory (KBCI); Post-traumatic Stress Disorder Checklist for DSM-5 (PCL-5); Patient Health Questionnaire (PHQ-9); Veterans RAND 36 Item Health Survey (VR-36); Epworth Sleepiness Scale (ESS); Feasibility of Intervention Measure (FIM)/Intervention Appropriateness Measure (IAM)/Acceptability of Intervention Measure (AIM); Self Efficacy for Symptom Management (SESx); NIH Toolbox - cognition; Memory Complaints Inventory (MCI); Inventory of Problems (IOP)
Supporting Information: CSR
Time Frame: Beginning after data collection ends with no end date
Access Criteria: Brain Injury Rehabilitation Service at Brooke Army Medical Center, Brain Injury Rehabilitation Service at Desmond T. Doss Health Clinic and McMaster University will be sent de-identified data that will be transmitted using DoD SAFE, which is a DoD endorsed platform for transferring data securely; De-identified data will be uploaded directly to Federal Interagency Traumatic Brain Injury Research (FITBIR) database;

REFERENCES:
- [Background] Cicerone KD, Azulay J. Perceived self-efficacy and life satisfaction after traumatic brain injury. J Head Trauma Rehabil. 2007 Sep-Oct;22(5):257-66. doi: 10.1097/01.HTR.0000290970.56130.81. PMID 17878767
- [Background] Corrigan JD, Bogner J. Initial reliability and validity of the Ohio State University TBI Identification Method. J Head Trauma Rehabil. 2007 Nov-Dec;22(6):318-29. doi: 10.1097/01.HTR.0000300227.67748.77. PMID 18025964
- [Background] Scheffler B, Schimbock F, Scholer A, Rosner K, Spallek J, Kopkow C. Tailored GuideLine Implementation in STrokE Rehabilitation (GLISTER) in Germany. Protocol of a Mixed Methods Study Using the Behavior Change Wheel and the Theoretical Domains Framework. Front Neurol. 2022 Jul 27;13:828521. doi: 10.3389/fneur.2022.828521. eCollection 2022. PMID 35968277
- [Background] Gromatsky M, Sullivan SR, Mitchell EL, Spears AP, Edwards ER, Goodman M. Feasibility and acceptability of VA CONNECT: Caring for our nation's needs electronically during the COVID-19 transition. Psychiatry Res. 2021 Feb;296:113700. doi: 10.1016/j.psychres.2020.113700. Epub 2020 Dec 31. PMID 33422845
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Kendzerska TB, Smith PM, Brignardello-Petersen R, Leung RS, Tomlinson GA. Evaluation of the measurement properties of the Epworth sleepiness scale: a systematic review. Sleep Med Rev. 2014 Aug;18(4):321-31. doi: 10.1016/j.smrv.2013.08.002. Epub 2013 Aug 22. PMID 24135493
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Kazis LE, Ren XS, Lee A, Skinner K, Rogers W, Clark J, Miller DR. Health status in VA patients: results from the Veterans Health Study. Am J Med Qual. 1999 Jan-Feb;14(1):28-38. doi: 10.1177/106286069901400105. PMID 10446661
- [Background] Beard C, Hsu KJ, Rifkin LS, Busch AB, Bjorgvinsson T. Validation of the PHQ-9 in a psychiatric sample. J Affect Disord. 2016 Mar 15;193:267-73. doi: 10.1016/j.jad.2015.12.075. Epub 2015 Dec 31. PMID 26774513
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Clapp JD, Kemp JJ, Cox KS, Tuerk PW. PATTERNS OF CHANGE IN RESPONSE TO PROLONGED EXPOSURE: IMPLICATIONS FOR TREATMENT OUTCOME. Depress Anxiety. 2016 Sep;33(9):807-15. doi: 10.1002/da.22534. Epub 2016 Jun 20. PMID 27321062
- [Background] Wortmann JH, Jordan AH, Weathers FW, Resick PA, Dondanville KA, Hall-Clark B, Foa EB, Young-McCaughan S, Yarvis JS, Hembree EA, Mintz J, Peterson AL, Litz BT. Psychometric analysis of the PTSD Checklist-5 (PCL-5) among treatment-seeking military service members. Psychol Assess. 2016 Nov;28(11):1392-1403. doi: 10.1037/pas0000260. Epub 2016 Jan 11. PMID 26751087
- [Background] Bovin MJ, Marx BP, Weathers FW, Gallagher MW, Rodriguez P, Schnurr PP, Keane TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in veterans. Psychol Assess. 2016 Nov;28(11):1379-1391. doi: 10.1037/pas0000254. Epub 2015 Dec 14. PMID 26653052
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Vanderploeg RD, Belanger HG, Duchnick JD, Curtiss G. Awareness problems following moderate to severe traumatic brain injury: Prevalence, assessment methods, and injury correlates. J Rehabil Res Dev. 2007;44(7):937-50. doi: 10.1682/jrrd.2006.12.0163. PMID 18075951
- [Background] Kolitz BP, Vanderploeg RD, Curtiss G. Development of the Key Behaviors Change Inventory: a traumatic brain injury behavioral outcome assessment instrument. Arch Phys Med Rehabil. 2003 Feb;84(2):277-84. doi: 10.1053/apmr.2003.50100. PMID 12601661
- [Background] Hoover PJ, Nix CA, Llop JZ, Lu LH, Bowles AO, Caban JJ. Correlations Between the Neurobehavioral Symptom Inventory and Other Commonly Used Questionnaires for Traumatic Brain Injury. Mil Med. 2023 Jul 22;188(7-8):usab559. doi: 10.1093/milmed/usab559. Epub 2022 Jan 12. PMID 35023563
- [Background] King PR, Donnelly KT, Donnelly JP, Dunnam M, Warner G, Kittleson CJ, Bradshaw CB, Alt M, Meier ST. Psychometric study of the Neurobehavioral Symptom Inventory. J Rehabil Res Dev. 2012;49(6):879-88. doi: 10.1682/jrrd.2011.03.0051. PMID 23299259
- [Background] Meterko M, Baker E, Stolzmann KL, Hendricks AM, Cicerone KD, Lew HL. Psychometric assessment of the Neurobehavioral Symptom Inventory-22: the structure of persistent postconcussive symptoms following deployment-related mild traumatic brain injury among veterans. J Head Trauma Rehabil. 2012 Jan-Feb;27(1):55-62. doi: 10.1097/HTR.0b013e318230fb17. No abstract available. PMID 22190009
- [Background] Vanderploeg RD, Silva MA, Soble JR, Curtiss G, Belanger HG, Donnell AJ, Scott SG. The structure of postconcussion symptoms on the Neurobehavioral Symptom Inventory: a comparison of alternative models. J Head Trauma Rehabil. 2015 Jan-Feb;30(1):1-11. doi: 10.1097/HTR.0000000000000009. PMID 24263177
- [Background] Vanderploeg RD, Cooper DB, Belanger HG, Donnell AJ, Kennedy JE, Hopewell CA, Scott SG. Screening for postdeployment conditions: development and cross-validation of an embedded validity scale in the neurobehavioral symptom inventory. J Head Trauma Rehabil. 2014 Jan-Feb;29(1):1-10. doi: 10.1097/HTR.0b013e318281966e. PMID 23474880
- [Background] Hardin KY, Black C, Caldbick K, Kelly M, Malhotra A, Tidd C, Vallentin T, Turkstra LS. Current Practices Among Speech-Language Pathologists for Mild Traumatic Brain Injury: A Mixed-Methods Modified Delphi Approach. Am J Speech Lang Pathol. 2021 Jul 14;30(4):1625-1655. doi: 10.1044/2021_AJSLP-20-00311. Epub 2021 May 26. PMID 34038183
- [Background] Malec JF, Smigielski JS, DePompolo RW. Goal attainment scaling and outcome measurement in postacute brain injury rehabilitation. Arch Phys Med Rehabil. 1991 Feb;72(2):138-43. PMID 1991015
- [Background] Geusgens CA, Winkens I, van Heugten CM, Jolles J, van den Heuvel WJ. Occurrence and measurement of transfer in cognitive rehabilitation: A critical review. J Rehabil Med. 2007 Jul;39(6):425-39. doi: 10.2340/16501977-0092. PMID 17624476
- [Background] Dunlosky J, Rawson KA, Marsh EJ, Nathan MJ, Willingham DT. Improving Students' Learning With Effective Learning Techniques: Promising Directions From Cognitive and Educational Psychology. Psychol Sci Public Interest. 2013 Jan;14(1):4-58. doi: 10.1177/1529100612453266. PMID 26173288
- [Background] Van Stan JH, Holmes J, Wengerd L, Juckett LA, Whyte J, Pinto SM, Katz LW, Wolfberg J. Rehabilitation Treatment Specification System: Identifying Barriers, Facilitators, and Strategies for Implementation in Research, Education, and Clinical Care. Arch Phys Med Rehabil. 2023 Apr;104(4):562-568. doi: 10.1016/j.apmr.2022.09.021. Epub 2022 Oct 26. PMID 36306923
- [Background] Meulenbroek P, Ness B, Lemoncello R, Byom L, MacDonald S, O'Neil-Pirozzi TM, Moore Sohlberg M. Social communication following traumatic brain injury part 2: Identifying effective treatment ingredients. Int J Speech Lang Pathol. 2019 Apr;21(2):128-142. doi: 10.1080/17549507.2019.1583281. Epub 2019 Apr 8. PMID 30955383
- [Background] Sikkes SAM, Tang Y, Jutten RJ, Wesselman LMP, Turkstra LS, Brodaty H, Clare L, Cassidy-Eagle E, Cox KL, Chetelat G, Dautricourt S, Dhana K, Dodge H, Droes RM, Hampstead BM, Holland T, Lampit A, Laver K, Lutz A, Lautenschlager NT, McCurry SM, Meiland FJM, Morris MC, Mueller KD, Peters R, Ridel G, Spector A, van der Steen JT, Tamplin J, Thompson Z; ISTAART Non-pharmacological Interventions Professional Interest Area; Bahar-Fuchs A. Toward a theory-based specification of non-pharmacological treatments in aging and dementia: Focused reviews and methodological recommendations. Alzheimers Dement. 2021 Feb;17(2):255-270. doi: 10.1002/alz.12188. Epub 2020 Nov 20. PMID 33215876
- [Background] Kinney AR, Middleton A, Graham JE. Evaluating the Strength of Evidence in Favor of Rehabilitation Effects: A Bayesian Analysis. Ann Phys Rehabil Med. 2022 Jan;65(1):101503. doi: 10.1016/j.rehab.2021.101503. Epub 2021 Nov 14. PMID 33667720
- [Background] Venkatesan UM, Ramanathan-Elion DM. Psychoeducation as Precision Health in Military-Related Mild Traumatic Brain Injury. Arch Phys Med Rehabil. 2022 Jun;103(6):1222-1232. doi: 10.1016/j.apmr.2021.08.012. Epub 2021 Sep 10. PMID 34516996
- [Background] Helou LB, Gartner-Schmidt JL, Hapner ER, Schneider SL, Van Stan JH. Mapping Meta-Therapy in Voice Interventions onto the Rehabilitation Treatment Specification System. Semin Speech Lang. 2021 Jan;42(1):5-18. doi: 10.1055/s-0040-1722756. Epub 2021 Feb 17. PMID 33596600
- [Background] Basilakos A, Hula WD, Johnson LP, Kiran S, Walker GM, Fridriksson J. Defining the Neurobiological Mechanisms of Action in Aphasia Therapies: Applying the Rehabilitation Treatment Specification System Framework to Research and Practice in Aphasia. Arch Phys Med Rehabil. 2022 Mar;103(3):581-589. doi: 10.1016/j.apmr.2021.10.017. Epub 2021 Nov 5. PMID 34748759
- [Background] Belanger HG, Vanderploeg RD, Curtiss G, Armistead-Jehle P, Kennedy JE, Tate DF, Eapen BC, Bowles AO, Cooper DB. Self-efficacy predicts response to cognitive rehabilitation in military service members with post-concussive symptoms. Neuropsychol Rehabil. 2020 Jul;30(6):1190-1203. doi: 10.1080/09602011.2019.1575245. Epub 2019 Feb 15. PMID 30764711
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Dejong G, Horn SD, Gassaway JA, Slavin MD, Dijkers MP. Toward a taxonomy of rehabilitation interventions: Using an inductive approach to examine the "black box" of rehabilitation. Arch Phys Med Rehabil. 2004 Apr;85(4):678-86. doi: 10.1016/j.apmr.2003.06.033. PMID 15083447
- [Background] Whyte J. Contributions of treatment theory and enablement theory to rehabilitation research and practice. Arch Phys Med Rehabil. 2014 Jan;95(1 Suppl):S17-23.e2. doi: 10.1016/j.apmr.2013.02.029. PMID 24370321
- [Background] Boutron I, Altman DG, Moher D, Schulz KF, Ravaud P; CONSORT NPT Group. CONSORT Statement for Randomized Trials of Nonpharmacologic Treatments: A 2017 Update and a CONSORT Extension for Nonpharmacologic Trial Abstracts. Ann Intern Med. 2017 Jul 4;167(1):40-47. doi: 10.7326/M17-0046. Epub 2017 Jun 20. PMID 28630973
- [Background] Hart T, Dijkers MP, Whyte J, Turkstra LS, Zanca JM, Packel A, Van Stan JH, Ferraro M, Chen C. A Theory-Driven System for the Specification of Rehabilitation Treatments. Arch Phys Med Rehabil. 2019 Jan;100(1):172-180. doi: 10.1016/j.apmr.2018.09.109. Epub 2018 Sep 27. PMID 30267669
- [Background] Hart T, Tsaousides T, Zanca JM, Whyte J, Packel A, Ferraro M, Dijkers MP. Toward a theory-driven classification of rehabilitation treatments. Arch Phys Med Rehabil. 2014 Jan;95(1 Suppl):S33-44.e2. doi: 10.1016/j.apmr.2013.05.032. PMID 24370323
- [Background] Turkstra LS, Norman R, Whyte J, Dijkers MP, Hart T. Knowing What We're Doing: Why Specification of Treatment Methods Is Critical for Evidence-Based Practice in Speech-Language Pathology. Am J Speech Lang Pathol. 2016 May 1;25(2):164-71. doi: 10.1044/2015_AJSLP-15-0060. PMID 27145191
- [Background] Fure SCR, Howe EI, Andelic N, Brunborg C, Sveen U, Roe C, Rike PO, Olsen A, Spjelkavik O, Ugelstad H, Lu J, Ponsford J, Twamley EW, Hellstrom T, Lovstad M. Cognitive and vocational rehabilitation after mild-to-moderate traumatic brain injury: A randomised controlled trial. Ann Phys Rehabil Med. 2021 Sep;64(5):101538. doi: 10.1016/j.rehab.2021.101538. Epub 2021 Jul 22. PMID 33957293
- [Background] Samuelson KW, Engle K, Abadjian L, Jordan J, Bartel A, Talbot M, Powers T, Bryan L, Benight C. Cognitive Training for Mild Traumatic Brain Injury and Posttraumatic Stress Disorder. Front Neurol. 2020 Nov 26;11:569005. doi: 10.3389/fneur.2020.569005. eCollection 2020. PMID 33324318
- [Background] Mahncke HW, DeGutis J, Levin H, Newsome MR, Bell MD, Grills C, French LM, Sullivan KW, Kim SJ, Rose A, Stasio C, Merzenich MM. A randomized clinical trial of plasticity-based cognitive training in mild traumatic brain injury. Brain. 2021 Aug 17;144(7):1994-2008. doi: 10.1093/brain/awab202. PMID 34312662
- [Background] Storzbach D, Twamley EW, Roost MS, Golshan S, Williams RM, O'Neil M, Jak AJ, Turner AP, Kowalski HM, Pagulayan KF, Huckans M. Compensatory Cognitive Training for Operation Enduring Freedom/Operation Iraqi Freedom/Operation New Dawn Veterans With Mild Traumatic Brain Injury. J Head Trauma Rehabil. 2017 Jan/Feb;32(1):16-24. doi: 10.1097/HTR.0000000000000228. PMID 27022961
- [Background] Kennedy JE, Cooper DB, Curtiss G, Shelton JL, Bowles AO, Tate DF, Eapen BC, Vanderploeg RD. Research Letter: Long-Term Outcomes Following Cognitive Rehabilitation for Mild Traumatic Brain Injury: A 5-Year Follow-Up of a Cohort From the SCORE Randomized Clinical Trial. J Head Trauma Rehabil. 2022 Nov-Dec 01;37(6):390-395. doi: 10.1097/HTR.0000000000000800. Epub 2022 Jul 20. PMID 35862897
- [Background] Fetta J, Starkweather A, Gill JM. Computer-Based Cognitive Rehabilitation Interventions for Traumatic Brain Injury: A Critical Review of the Literature. J Neurosci Nurs. 2017 Aug;49(4):235-240. doi: 10.1097/JNN.0000000000000298. PMID 28661947
- [Background] Cooper DB, Bunner AE, Kennedy JE, Balldin V, Tate DF, Eapen BC, Jaramillo CA. Treatment of persistent post-concussive symptoms after mild traumatic brain injury: a systematic review of cognitive rehabilitation and behavioral health interventions in military service members and veterans. Brain Imaging Behav. 2015 Sep;9(3):403-20. doi: 10.1007/s11682-015-9440-2. PMID 26330376
- [Background] Borg J, Holm L, Peloso PM, Cassidy JD, Carroll LJ, von Holst H, Paniak C, Yates D; WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. Non-surgical intervention and cost for mild traumatic brain injury: results of the WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. J Rehabil Med. 2004 Feb;(43 Suppl):76-83. doi: 10.1080/16501960410023840. PMID 15083872
- [Background] Carroll LJ, Cassidy JD, Holm L, Kraus J, Coronado VG; WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. Methodological issues and research recommendations for mild traumatic brain injury: the WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. J Rehabil Med. 2004 Feb;(43 Suppl):113-25. doi: 10.1080/16501960410023877. PMID 15083875
- [Background] Rosenthal M. Mild traumatic brain injury syndrome. Ann Emerg Med. 1993 Jun;22(6):1048-51. doi: 10.1016/s0196-0644(05)82749-0. PMID 8503524
- [Background] Cooper DB, Bowles AO, Kennedy JE, Curtiss G, French LM, Tate DF, Vanderploeg RD. Cognitive Rehabilitation for Military Service Members With Mild Traumatic Brain Injury: A Randomized Clinical Trial. J Head Trauma Rehabil. 2017 May/Jun;32(3):E1-E15. doi: 10.1097/HTR.0000000000000254. PMID 27603763
- [Background] Klein OA, Drummond A, Mhizha-Murira JR, Mansford L, dasNair R. Effectiveness of cognitive rehabilitation for people with multiple sclerosis: a meta-synthesis of patient perspectives. Neuropsychol Rehabil. 2019 May;29(4):491-512. doi: 10.1080/09602011.2017.1309323. Epub 2017 May 1. PMID 28457198
- [Background] Resch C, Rosema S, Hurks P, de Kloet A, van Heugten C. Searching for effective components of cognitive rehabilitation for children and adolescents with acquired brain injury: A systematic review. Brain Inj. 2018;32(6):679-692. doi: 10.1080/02699052.2018.1458335. Epub 2018 Apr 5. PMID 29621405
- [Background] Seal KH, Bertenthal D, Barnes DE, Byers AL, Strigo I, Yaffe K; Chronic Effects of Neurotrauma Consortium Study Group. Association of Traumatic Brain Injury With Chronic Pain in Iraq and Afghanistan Veterans: Effect of Comorbid Mental Health Conditions. Arch Phys Med Rehabil. 2017 Aug;98(8):1636-1645. doi: 10.1016/j.apmr.2017.03.026. Epub 2017 Apr 25. PMID 28455190
- [Background] Walker WC, Hirsch S, Carne W, Nolen T, Cifu DX, Wilde EA, Levin HS, Brearly TW, Eapen BC, Williams R. Chronic Effects of Neurotrauma Consortium (CENC) multicentre study interim analysis: Differences between participants with positive versus negative mild TBI histories. Brain Inj. 2018;32(9):1079-1089. doi: 10.1080/02699052.2018.1479041. Epub 2018 May 31. PMID 29851515
- [Background] Martindale SL, Farrell-Carnahan LV, Ulmer CS, Kimbrel NA, McDonald SD, Rowland JA; VA Mid-Atlantic MIRECC Registry Workgroup. Sleep quality in returning veterans: The influence of mild traumatic brain injury. Rehabil Psychol. 2017 Nov;62(4):563-570. doi: 10.1037/rep0000159. Epub 2017 Jul 13. PMID 28703617
- [Background] Soble JR, Silva MA, Vanderploeg RD, Curtiss G, Belanger HG, Donnell AJ, Scott SG. Normative Data for the Neurobehavioral Symptom Inventory (NSI) and post-concussion symptom profiles among TBI, PTSD, and nonclinical samples. Clin Neuropsychol. 2014;28(4):614-32. doi: 10.1080/13854046.2014.894576. Epub 2014 Mar 14. PMID 24625213
- [Background] Lange RT, Lippa SM, French LM, Bailie JM, Gartner RL, Driscoll AE, Wright MM, Sullivan JK, Varbedian NV, Barnhart EA, Holzinger JB, Schaper AL, Reese MA, Brandler BJ, Camelo-Lopez V, Brickell TA. Long-term neurobehavioural symptom reporting following mild, moderate, severe, and penetrating traumatic brain injury in U.S. military service members. Neuropsychol Rehabil. 2020 Oct;30(9):1762-1785. doi: 10.1080/09602011.2019.1604385. Epub 2019 Apr 19. PMID 31003592
- See also: DOD TBI Worldwide Numbers — https://health.mil/Military-Health-Topics/Centers-of-Excellence/Traumatic-Brain-Injury-Center-of-Excellence/DOD-TBI-Worldwide-Numbers
- See also: VA/DoD Clinical Practice Guideline for the Management and Rehabilitation of Post-Acute Mild Traumatic Brain Injury — https://www.healthquality.va.gov/guidelines/rehab/mtbi/
- See also: International Classification of Health Interventions (ICHI) — https://www.who.int/classifications/international-classification-of-health-interventions
- See also: NIH Toolbox Cognition Battery — https://nihtoolbox.org/domain/cognition/